CLINICAL TRIAL: NCT01215318
Title: Source and Prevention of Urinary Contamination of Vaginal Tampons During 18F-2-fluoro-2-deoxy-D-glucose (FDG) Positron Emission Tomography (PET) Examinations
Brief Title: FDG Uptake in Vaginal Tampons is Due to Urine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Irene Burger (Other)
Responsible Party: Sponsor-Investigator, Irene Burger, Attending physician, University of Zurich
Organization: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: KEK-ZH-NR: 2010-0014
Record Dates: First submitted 2010-10-04; First posted 2010-10-06 (Estimated); Results first posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Cancer
Keywords: FDG PET/CT, vaginal tampon, urinary contamination, pitfall
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: randomly assigned to either modified or unmodified tampons
Oversight: Data Monitoring Committee: No

ARMS (2):
- Modified vaginal tampons (Experimental): Patients using modified vaginal tampons during FDG PET/CT
  Interventions: Device: modified vaginal tampon
- Unmodified vaginal tampons (Placebo Comparator): Patients using unmodified vaginal tampons during FDG PET/CT
  Interventions: Device: modified vaginal tampon

INTERVENTIONS:
Device: modified vaginal tampon — modified vaginal tampons versus unmodified vaginal tampons, comparing the urinary contamination
  Other Names: Ob® Regular; Johnson & Johnson, with silicon seal

SUMMARY:
The etiology of FDG uptake in vaginal tampons during PET/CT examinations remains unclear and can potentially impair image interpretation.

The aim of this study is to determine the etiology of this artefact and identify potential means how to prevent it.

DETAILED DESCRIPTION:
In this prospective, Institutional Review board approved study we included 44 women referred to FDG PET/CT for staging or follow-up in an oncology setting. All women were provided a normal commercial or modified vaginal tampon with a silicon coated base to be used during examination. Images were analyzed to determine the localization and the FDG uptake in the tampons. Between the uptake phase and imaging, all patients were asked to void. After image acquisition, tampons were individually analyzed for creatinine concentration, blood traces, position relative to the pubococcygeal line, and FDG activity. Statistical significance was determined by means of the Mann-Whitney U test.

ELIGIBILITY:
Inclusion criteria: premenopausal women with known or suspected malignancies who regularly used vaginal tampons during menstruation and thus were familiar with their use

Exclusion criteria: No cervical or genital carcinoma. No vaginal infection.

Ages: 20 Years to 48 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2010-02-02 (Actual); Primary Completion 2010-08-02 (Actual); Study Completion 2010-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Premenopausal women referred for FDG PET/CT examination for staging or follow up of malign disease, were given a modified or unmodified vaginal tampon during the PET/CT examination.
Pre-assignment Details: Women with urogenital carcinoma were excluded.
Groups:
- Modified Vaginal Tampons: Patients wearing modified tampons during PET/CT
- Unmodified Vaginal Tampons: Patients wearing unmodified vaginal tampons during FDG PET/CT
Period: Overall Study
Arm/Group | Modified Vaginal Tampons | Unmodified Vaginal Tampons
Started | 20 | 24
Completed | 20 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Modified Vaginal Tampons: Patients wearing modified vaginal tampons during PET/CT
- Unmodified Vaginal Tampons: Patients wearing unmodified vaginal tampons during PET/CT
- Total: Total of all reporting groups
Arm/Group | Modified Vaginal Tampons | Unmodified Vaginal Tampons | Total
Number analyzed (Participants) | 20 | 24 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 24 | 44
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (7.7) | 37 (8.4) | 39 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 24 | 44
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 20 | 24 | 44

OUTCOME MEASURES:

1. Primary Outcome: Number of FDG Positive Tampoons
Description: Number of FDG positive Tampoons with an SUV > 3
Time Frame: 1 month
Measure: Number; unit: FDG positive tampons
Units Other Than Participants: vaginal tampons
Groups:
- Modified Vaginal Tampons: Patients wearing modified tampons during FDG PET/CT
- Unmodified Vaginal Tampons: Patients wearing unmodified tampons during FDG PET/CT
Arm/Group | Modified Vaginal Tampons | Unmodified Vaginal Tampons
Number analyzed (Participants) | 20 | 24
Number analyzed (vaginal tampons) | 20 | 24
FDG positive tampons | 2 | 10

2. Secondary Outcome: Tampon Position Relative to the Pubococcygeal Line
Description: measure tampon position in regard to the pubococcygeal line to identify if positioning is responsible for urinary contamination.
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: vaginal tampons
Groups:
- Modified Vaginal Tampons; Unmodified Vaginal Tampons: Patients wearing modified vaginal tampon during PET/CT
Arm/Group | Modified Vaginal Tampons | Unmodified Vaginal Tampons
Number analyzed (Participants) | 20 | 24
Number analyzed (vaginal tampons) | 20 | 24
mm | 5.9 (17) | 5.1 (11)

ADVERSE EVENTS:
Time Frame: During FDG PET/CT scan (2 hours)
Description: Dyscomfort
Groups:
- Unmodified Vaginal Tampons: Patients wearing unmodified vaginal tampon during PET/CT
Arm/Group | Modified Vaginal Tampons | Unmodified Vaginal Tampons
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/24
Other Adverse Events (participants affected / at risk) | 0/20 | 0/24

LIMITATIONS AND CAVEATS:
absence of gynecological examination. Vaginal tampon position was only assessed with respect to the pubococcygeal line visualized on computer tomography.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No